CLINICAL TRIAL: NCT04829877
Title: Trajectory of Psychological Distress Among Infertility Women: Efficacy and Mechanism of Mind-body Intervention With Heart Rate Variability Biofeedback
Brief Title: Trajectory of Psychological Distress Among Infertility Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University (Other)
Responsible Party: Principal Investigator, Shu Yu Kuo, Principal investigator, Taipei Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: N201807030
Record Dates: First submitted 2021-03-31; First posted 2021-04-02 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Infertility; Heart Rate Variability; Biofeedback
Keywords: infertility; mind-body intervention; heart rate variability; biofeedback; psychological distress
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Web-based mind-body intervention with HRVB (Experimental): Both standard usual care and the web-based mind-body intervention with HRV biofeedback (MBI-HRVB) will be provided to the participants. The web-based mind-body intervention with HRV biofeedback program consisted of 5-week training sessions and breathing training.
  Interventions: Behavioral: Web-based mind-body intervention with HRVB
- Web-based mind-body intervention (Experimental): Both standard usual care and the web-based mind-body intervention will be provided to the participants. The web-based mind-body intervention program consisted of 5-week training sessions.
  Interventions: Behavioral: Web-based mind-body intervention
- Control (No Intervention): The women in the control group will receive the standard usual care provided at the fertility clinic. The standard care protocols encompass elements such as routine assessment and health education at each visit. Participants enrolled in the control group will be approached once a week by a nurse to provide health consultation about fertility treatment, medication, signs, and symptoms of discomfort for five weeks.

INTERVENTIONS:
Behavioral: Web-based mind-body intervention with HRVB — The web-based mind-body intervention with HRVB contains the following components: 1) Breathing training with HRV biofeedback; 2) 5 different topics will be included ; 3) Home exercise of slow breathing and mindfulness exercise.
  Arms: Web-based mind-body intervention with HRVB
Behavioral: Web-based mind-body intervention — The web-based mind-body intervention will receive 5 different topics courses.
  Arms: Web-based mind-body intervention

SUMMARY:
Background: Infertility is a serious reproductive health issue and affects 48.5 million couples worldwide. Women undergoing fertility treatment often experienced psychological distress but also social stigma that is close linked to later pregnancy outcome. Despite the advancement in assisted reproductive technology, effective interventions for reducing stress, anxiety, and depressive symptoms for infertility women remain lacking.

Objectives: The objective of this proposal is to evaluate the efficacy of web-based mind-body intervention combining HRV biofeedback on the infertility women's anxiety symptoms, levels of depression, HRV function, mindful awareness, infertility self-efficacy, and pregnancy rates.

Methods: We plan to conduct a randomized controlled trial on the web-based mind-body intervention combining heart rate variability biofeedback. Eligible women will be recruited and randomized into three groups. Intention-to-treat analysis and mixed regression modeling will be used to estimate the effectiveness of the interventions.

Anticipatory results: Effective strategies will be determined for infertility women.

DETAILED DESCRIPTION:
A designed data entry system for the current study will be developed to ensure an error-proof process. It is important to inspect data for outliers, wild code, and consistency to maintain the data quality in the pre-analysis data phase. We will assess the amount and pattern of missing values by using descriptive statistics, such as frequency and percentage. The pattern of missing data will be identified and decide whether the missing completely at random or not. The appropriate corresponding method will be adopted for the subsequent statistical analyses. For example, the mean imputation is considered when the percentage of items missing at a given questionnaire is less than 10 %. The mean imputation will be used to replaces a missing value with the item mean when applicable. The comparison between complete case analysis and imputation data will be performed to assess the reliability and validity of the results.

ELIGIBILITY:
Inclusion Criteria:

* 20-year-old and above
* Seeking infertility care
* Contemplating pregnancy
* Intended to start their ART cycle
* Able to speak Taiwanese or Mandarin

Exclusion Criteria:

* Diagnosis of cardiovascular disease, depressive disorder, anxiety disorder, cardiac arrhythmia
* Already had started their ART treatment
* Taking medications that might affect ANS activity

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 750 (Estimated)
Dates: Start 2022-04-19 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Anxiety | Baseline
  Anxiety symptoms will be assessed using the Taiwanese version of the State Anxiety Inventory (SAI).
Anxiety | 1 week post-intervention
  Anxiety symptoms will be assessed using the Taiwanese version of the State Anxiety Inventory (SAI).
Anxiety | 1 month post-intervention
  Anxiety symptoms will be assessed using the Taiwanese version of the State Anxiety Inventory (SAI).
Anxiety | 2 month post-intervention
  Anxiety symptoms will be assessed using the Taiwanese version of the State Anxiety Inventory (SAI).
Anxiety | 3 month post-intervention
  Anxiety symptoms will be assessed using the Taiwanese version of the State Anxiety Inventory (SAI).

SECONDARY OUTCOMES:
Depressive symptoms | Baseline, post-intervention 1 week, month 1 , 2 and 3
  The Taiwanese version of the Beck Depression Inventory (BDI) will be used to assess depressive symptoms among infertility women.
HRV function | Baseline, post-intervention 1 week, month 1 , 2 and 3
  The HRV signal will be measured using standard equipment.
Mindful awareness | Baseline, post-intervention 1 week, month 1 , 2 and 3
  The Taiwanese version of the Five Facet Mindfulness Questionnaire (FFMQ) will be adopted to assess levels of mindfulness.
Infertility self-efficacy | Baseline, post-intervention 1 week, month 1 , 2 and 3
  The infertility Self-Efficacy Scale (ISE) will be used for studied women.
Pregnancy rates | 15 days after embryo transfer or ultrasound
  Clinical pregnancy will be defined as a positive blood, urinary pregnancy test.

CONTACTS AND LOCATIONS:
Overall Officials: Shu-Yu Kuo, Phd, Principal Investigator — Taipei Medical University
Locations (1):
- Infertility clinic, Taipei, Taiwan